CLINICAL TRIAL: NCT02979275
Title: Correlation of Brain and Thenar Muscle Oximetry During Cardiac Surgery With Parameters of Acute Kidney Injury in Adult Cardiac Surgical Patients Operated on Cardiopulmonary Bypass
Brief Title: Correlation of Brain and Thenar Muscle Oximetry During Cardiac Surgery With Parameters of Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Romuald Lango, Dr hab. med. Romuald Lango, Medical University of Gdansk
Other Study IDs: NKEBN/122/2014; grant ST-44 (Other Grant/Funding Number: Medical University of Gdansk)
Record Dates: First submitted 2016-11-21; First posted 2016-12-01 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury; Heart Valve Diseases
Keywords: acute kidney injury; cardiopulmonary bypass; neutrophil gelatinase-associated lipocalin; tissue hypoxia
MeSH Terms: conditions — Acute Kidney Injury; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from blood samples obtained at 10 timepoints before, during, and after the cardiac surgical operation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BRAIN+THENAR MUSCLE INVOS: Patients undergoing open heart surgery on cardiopulmonary bypass.
  Interventions: Procedure: Open heart surgery on cardiopulmonary bypass.

INTERVENTIONS:
Procedure: Open heart surgery on cardiopulmonary bypass. — Brain oximetry and tissue saturation will be measured during operation. NGAL, cystatin-C, and Acute Kidney Injury Network (AKIN) criteria of AKI will be assessed durin first post-op day.

SUMMARY:
Identification of risk factors of acute kidney injury (AKI). It is hypothesized that there might be a correlation between brain oximetry, tissue saturation of thenar muscle and marker of AKI in blood - neutrophil gelatinase-associated lipocalin (NGAL) - measured in blood samples during the first post-op day.

DETAILED DESCRIPTION:
The day before operation, after verification of inclusion and exclusion criteria, the visiting anesthesiologist will explain to the patient the aim of the study. By signing an informed consent the patient will be recruited into the study. On the evening before operation the patient will receive the statin in a dose taken along.

In the OR the anesthesiologist will verify if creatinin and blood urea nitrogen were measured the day before operation - if not, a blood sample for the test will be obtained and sent to perform the tests.

Before induction of anesthesia a bi-spectral index (BIS) probe will be placed on the patients forehead. Above the BIS probe a INVOS(TM) probe for brain oximetry (5100 C Cerebral/Somatic Oximeter, Somanetics, Medtronic) will be placed.

Brain oximetry by near infrared saturation (NIRS) and tissue saturation on thenar muscle will be recorded before and during operation on nine timepoints.

As NIRS and thenar muscle saturation are non-routine non-invasive methods of intraoperative monitoring, patient had to sign an informed consent to participate into the study, and ethic committee approval for the study protocol was appealed and granted.

General anesthesia will be induced by: fentanyl 0.2 mg, propofol 0.5-1.5 mg/kg in bolus 200ml/godz.; and rocuronium - 0.5 mg/kg. After induction dexamethasone will be given in a dose of 0,7-1 mg/kg. For conduction of anesthesia before cardiopulmonary bypass (CPB) sevoflurane will be added to the inhaled mixture of air and oxygen. On CPB propofol will be given iv. In case of hemodynamic instability after commencing CPB, which will require catecholamines in a cumulative dose of > 1.5 standard, or in case of trouble to commence CPB, propofol will be replaced by midazolam in a dose 0.2-0.3 mg/kg/hour.

During anesthesia, first post-operative day and hospital stay a total of 278 variables will be recorded: hemodynamic parameters, iv fluid doses, inotropes, vasopressors, diuretics, urine output, transfusions, etc.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* signed informed consent
* scheduled for elective on-bypass cardiac surgery (aortic valve surgery, mitral valve surgery with/without tricuspid valve surgery, ascending aorta surgery with/without aortic valve surgery).

Exclusion Criteria:

* chronic kidney insufficiency (serum creatinine >2 mg/dL)
* active infection (i.e.: endocarditis)
* shock or tissue hypoperfusion before operation (blood lactate >3 mmol/L)
* left ventricle ejection fraction <25%
* vancomycin used for infection prophylaxis (i.e.: in immunosuppressed patients)
* history of ischaemic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patient scheduled for elective on-bypass cardiac surgery (aortic valve surgery, mitral valve surgery with/without tricuspid valve surgery, ascending aorta surgery with/without aortic valve surgery).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
NGAL | 3 hours after operation
  neutrophil gelatinase-associated lipocalin (NGAL) measured in blood samples

SECONDARY OUTCOMES:
NGAL on second day | second post-op day morning
  neutrophil gelatinase-associated lipocalin (NGAL) measured in blood samples
Cystatin C | second post-op day morning
  Cystatin-C measured in blood samples
Serum creatinine | second post-op day morning
  Serum creatinine in serum
Acute renal failure | 30 day / any time after operation before discharge from hospital
  Acute renal failure requiring renal replacement therapy or AKIN stage 3
In hospital mortality | 30 day / any time after operation before discharge from hospital
  Death from any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Lango, M.D., Ph.D., Study Director — Medical University of Gdańsk, Department of Cardiac Anesthesiology
Locations (1):
- Medical University of Gdańsk, Department of Cardiac Anesthesiology, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) may be done available to other researchers upon reasonable request directed to study director.